CLINICAL TRIAL: NCT01471990
Title: The Effect of PACAP38 and VIP on Migraine Patients Assessed by a 3-Tesla MR Scanner
Brief Title: Effect of PACAP38/VIP on Migraineurs Measured by Magnetic Resonance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Bispebjerg Hospital (Other); University Hospital, Gentofte, Copenhagen (Other); Lundbeck Foundation (Other); Cool Sorption Foundation of 1988 (Other)
Responsible Party: Principal Investigator, Faisal Mohammad Amin, medical doctor, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: H-1-2011-023
Record Dates: First submitted 2011-11-09; First posted 2011-11-16 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Migraine Without Aura
Keywords: PACAP38; MMA; migraine; angiography; VIP; vasodilatation
MeSH Terms: conditions — Migraine without Aura; Migraine Disorders; Aneurysm | interventions — Vasoactive Intestinal Peptide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PACAP38 (Active Comparator)
  Interventions: Drug: Pituitary Adenylate Cyclase-Activating Polypeptide-38
- VIP (Active Comparator)
  Interventions: Drug: Vasoactive Intestinal Peptide

INTERVENTIONS:
Drug: Pituitary Adenylate Cyclase-Activating Polypeptide-38 — 10 pmol/kg/min over 20 mins
  Arms: PACAP38
Drug: Vasoactive Intestinal Peptide — 8 pmol/kg/min over 20 mins
  Arms: VIP

SUMMARY:
The purpose of this study is to examine and compare the effect of pituitary adenylate cyclase-activating polypeptide-38 (PACAP38) and vasoactive intestinal polypeptide (VIP) on intracranial arteries and neuronal activity in patients with migraine without aura using a high resolution magnetic resonance imaging (MRI), including MR angiography (MRA) and functional MRI (fMRI).

MRA will be used to detect changes in intracranial artery circumferences before and after PACAP38 and VIP.

fMRI will be used oo detect changes in blood-oxygenation-level-dependent-signal (BOLD-signal).

PACAP38 but not VIP induces migraine like attacks in migraine patients. The migraine specific drug sumatriptan will be given to relieve pain and the effect will also be registered using MRA and fMRI.

ELIGIBILITY:
Inclusion Criteria:

* Healthy migraine patient without aura
* Age 18-40
* Weight 50-100 kg
* Fertile women must use safe contraceptives

Exclusion Criteria:

* Tension type headache more than 5 days per month
* Other primary headaches
* Daily use of medication except contraceptives
* Drug taken within 4 times the half life for the specific drug except contraceptives
* Pregnant or lactating women
* Exposure to radiation within the last year
* Hypotension or hypertension
* Cardiovascular or cerebrovascular disease
* Mental illness or substance abuse
* Other significant conditions determined by the examining doctor
* Contraindications to MRI scan
* Headache within the last 48 hours before start of trial

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Comparison between PACAP38 and VIP induced changes in intracranial artery circumference before and after infusions | Baseline, 20 minutes, 2 hours and 5 hours

SECONDARY OUTCOMES:
Headache scores | 24 hours
  hospital and post hospital phase
Comparison between PACAP38 and VIP induced changes in BOLD response | 5 hours
Change in intracranial artery circumference before and after injection of sumatriptan | 5 hours
Comparison between PACAP38 and VIP induced changes in brain structure | 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Amin, M.D., Principal Investigator — Danish Headache Centre and Department of Neurology, Glostrup Hospital, Faculty of Health Sciences, University of Copenhagen
Locations (1):
- Glostrup Hospital, Faculty of Health Sciences, University of Copenhagen, Glostrup Municipality, Denmark